CLINICAL TRIAL: NCT01150032
Title: Bone Quality and Improvement of Fracture Risk Prediction
Brief Title: Bone Quality Lyon Orleans
Acronym: QUALYOR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2009.588
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Osteopenic Women
Keywords: Osteoporosis; Fracture; Bone microarchitecture
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen plasma: for later genetic studies Frozen serum: for later studies on new potential marker of bone remodelling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteopenic women: Women with osteopenia: Bone Mineral Density T-score between -1.0 and -2.5 (for whom with clinical factor risk) or -3.0 (for whom without clinical factor risk)
  Interventions: Other: Bone quality complementary exams

INTERVENTIONS:
Other: Bone quality complementary exams — realisation of following exams to evaluate fracture risk in osteopenic women:
  * hip and wrist Dual energy X-ray Absorptiometry (DXA)
  * wrist and shin High-Resolution peripheral Quantitative Computed-Tomography(HR-pQCT)
  * hip Quantitative Computed Tomography (QCT)
  * High Resolution Digital X-Ray of calcaneum using BMA(tm) system
  * low-dose stereoradiography using EOS(tm) system (only for a sub-group of 60 voluntary subjects)

SUMMARY:
QUALYOR is a prospective study on the predictive value for fragility fracture of various new techniques assessing bone quality, among postmenopausal women with low bone mass.

ELIGIBILITY:
Inclusion Criteria:

* 50 or older women
* post-menopausal since at least one year
* with osteopenia (T-score between -1.0 and -2.5 (with clinical factor risk) or -3.0 (without clinical factor risk)

Exclusion Criteria:

* corticosteroid therapy > 3 months, at least 7.5mg/day equivalent prednisolon (stopped since at least 1 year)
* osteoporosis treatment antecedent
* fragility fracture antecedent
* on going post-menopausal hormonal treatment
* clinical signs of hepatic, cardiac or respiratory insufficiency, diseases possibly affecting bone metabolism
* life expectancy < 4 years, mental or serious illness

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 years old or older women with lowered Bone Mineral Density
Sampling Method: Non-Probability Sample
Enrollment: 1605 (Actual)
Dates: Start 2010-09-20 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Fragility fracture | 4 years
  Appearance of vertebral or non-vertebral fracture during the 4 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Roland CHAPURLAT, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier d'Orléans, Orléans

REFERENCES:
- [Derived] Chapurlat R, Pialat JB, Merle B, Confavreux E, Duvert F, Fontanges E, Khacef F, Peres SL, Schott AM, Lespessailles E. The QUALYOR (QUalite Osseuse LYon Orleans) study: a new cohort for non invasive evaluation of bone quality in postmenopausal osteoporosis. Rationale and study design. Arch Osteoporos. 2017 Dec 27;13(1):2. doi: 10.1007/s11657-017-0412-6. PMID 29282548